CLINICAL TRIAL: NCT03681405
Title: Support for Optimal Recovery Following Gynecologic Surgery Study (SOARING)
Brief Title: Supportive Programs for Supporting Optimal Recovery in Participants Undergoing Gynecological Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: IRB00052655; NCI-2018-01801 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 97218 (Other: Wake Forest University Health Sciences); P30CA012197 (NIH)
Record Dates: First submitted 2018-08-31; First posted 2018-09-24 (Actual); Results first posted 2021-06-24 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-11

CONDITIONS: Ovarian Neoplasm; Uterine Neoplasm
MeSH Terms: conditions — Ovarian Neoplasms; Uterine Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (eMMB) (Experimental): Participants will receive instruction on awareness meditation, breathing and relaxation, and awareness meditation. This will include a call with the interventionist to invite participants to initiate additional guidance upon request prior to surgery and a meeting by videoconferencing the day following surgery. Participants will also be given a self-directed video to be used before surgery and daily for two weeks following surgery.
  Interventions: Other: Informational Intervention; Other: Questionnaire Administration
- Group II (AC) (Active Comparator): Participants will receive caring attention. This will include a call with the interventionist to invite participants to initiate additional guidance upon request prior to surgery and a meeting by videoconferencing the day following surgery. Participants are also asked to write brief diary entries once before surgery and daily for two weeks following surgery.
  Interventions: Other: Questionnaire Administration; Behavioral: Telephone-Based Intervention

INTERVENTIONS:
Other: Informational Intervention — Given information about mindful movement and breathing
  Arms: Group I (eMMB)
Other: Questionnaire Administration — Ancillary studies
Behavioral: Telephone-Based Intervention — Receive caring attention phone call
  Arms: Group II (AC)

SUMMARY:
This trial studies how well two different supportive programs work in supporting optimal recovery in participants undergoing gynecological surgery. Supportive programs use different methods for helping participants cope with the surgical experience including gentle movements, counseling, writing, or relaxation techniques, and may help improve participants' well-being after gynecological surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To calculate recruitment, adherence, assessment completion, and retention rates.

SECONDARY OBJECTIVES:

I. Document the frequency of adverse events. II. Assess descriptive data on proposed outcomes (i.e., pain, sleep disturbances, psychological distress) for the next phase of study.) III. Qualitatively assess acceptability to guide future study planning.

OUTLINE: Participants are randomized to 1 of 2 groups.

GROUP I (MINDFUL MOVEMENT AND BREATHING [eMMB]): Participants will receive instruction on awareness meditation, breathing and relaxation, and awareness meditation. This will include a call with the interventionist to invite participants to initiate additional guidance upon request prior to surgery and a meeting by videoconferencing the day following surgery. Participants will also be given a self-directed video to be used before surgery and daily for two weeks following surgery.

GROUP II (ATTENTION CONTROL [AC]): Participants will receive caring attention. This will include a call with the interventionist to invite participants to initiate additional guidance upon request prior to surgery and a meeting by videoconferencing the day following surgery. Participants are also asked to write brief diary entries once before surgery and daily for two weeks following surgery.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for an abdominal gynecological surgery (i.e. uterine, ovarian) to remove a suspected malignancy.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of =< 1.
* Cognitively able to complete assessments as judged by the study team.
* Able to understand, read and write English.

Exclusion Criteria:

* Have schizophrenia or any other psychotic disorder.
* Have a diagnosed sleep disorder including untreated obstructive sleep apnea, periodic limb movement disorder, or restless leg syndrome.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-12-07 (Actual); Primary Completion 2020-04-09 (Actual); Study Completion 2020-04-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Sohl, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

REFERENCES:
- [Derived] Sohl SJ, Strahley AE, Tooze JA, Levine BJ, Kelly MG, Wheeler A, Evans S, Danhauer SC. Qualitative results from a randomized pilot study of eHealth Mindful Movement and Breathing to improve gynecologic cancer surgery outcomes. J Psychosoc Oncol. 2024;42(2):223-241. doi: 10.1080/07347332.2023.2236083. Epub 2023 Jul 18. PMID 37462260

RESULTS

PARTICIPANT FLOW:
Groups:
- Group I eHealth Mindful Movement and Breathing (eMMB): Participants will receive instruction on awareness meditation, breathing and relaxation, and awareness meditation. This will include a call with the interventionist to invite participants to initiate additional guidance upon request prior to surgery and a meeting by videoconferencing the day following surgery. Participants will also be given a self-directed video to be used before surgery and daily for two weeks following surgery.
  Informational Intervention: Given information about mindful movement and breathing
  Questionnaire Administration: Ancillary studies
- Group II Attention Control (AC): Participants will receive caring attention. This will include a call with the interventionist to invite participants to initiate additional guidance upon request prior to surgery and a meeting by videoconferencing the day following surgery. Participants are also asked to write brief diary entries once before surgery and daily for two weeks following surgery.
  Questionnaire Administration: Ancillary studies
  Telephone-Based Intervention: Receive caring attention phone call
Period: Overall Study
Arm/Group | Group I eHealth Mindful Movement and Breathing (eMMB) | Group II Attention Control (AC)
Started | 14 | 17
Completed | 13 | 17
Not Completed | 1 | 0
Not completed — Found to be ineligible after randomized | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group I (eMMB) | Group II (AC) | Total
Number analyzed (Participants) | 13 | 17 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.6 (13.0) | 58.9 (10.1) | 59.7 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 17 | 30
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 13 | 17 | 30
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 13 | 16 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 17 | 30

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Retained in the Study
Description: Will provide quantitative data to guide future study planning. Will calculate 95% confidence intervals for each of the feasibility measures to determine the range of estimates that are consistent with the data. Will track the number of screened participants, those who are eligible, and the percent who agree to participate. For those not meeting the eligibility criteria, reasons will be summarized. The proportion of participants and corresponding 95% CI for participants who participated in each group will be computed. Will use one-sample tests of binomial proportions to compare the recruitment, adherence, and retention rates to the hypothesized values of 50%, 70% and 70%, respectively.
Time Frame: Up to 2 weeks
Population: Of the 14 randomized to intervention for Group I, 1 person was removed from the study following randomization (and prior to filling out any surveys at baseline) due to ineligibility. For Group I and II, not all participants completed requirements of retention to be analyzed for the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants retained
Arm/Group | Group I (eMMB) | Group II (AC)
Number analyzed (Participants) | 14 | 17
percentage of participants retained | 78.6 [49.2 to 95.4] | 82.4 [56.6 to 96.2]

2. Primary Outcome: Percentage of Participants That Were Adhered to the Intervention
Description: Will provide quantitative data to guide future study planning. Will calculate 95% confidence intervals for each of the feasibility measures to determine the range of estimates that are consistent with the data. Will track the number of screened participants, those who are eligible, and the percent who agree to participate. For those not meeting the eligibility criteria, reasons will be summarized. The proportion of participants and corresponding 95% CI for participants who participated in each group will be computed.
Time Frame: Up to 5 weeks
Population: Of the 14 randomized to intervention for Group I, 1 person was removed from the study following randomization (and prior to filling out any surveys at baseline) due to ineligibility. For Group I and II, not all participants completed requirements of adherence to be analyzed for the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants adhered
Arm/Group | Group I (eMMB) | Group II (AC)
Number analyzed (Participants) | 14 | 17
percentage of participants adhered | 85.7 [57.2 to 98.2] | 70.6 [44.1 to 89.7]

3. Secondary Outcome: Change in Pain Intensity Per Patient Reported Outcomes Measurement Information System (PROMIS)
Description: Baseline analyses will include descriptive statistics of pain, background characteristics and other possible confounding variables by intervention group. The primary goal of the statistical analysis of these measures for this Aim will be to estimate standard deviations (SD) for use in future studies. A change in pain intensity between two or more time points (baseline, 2 weeks and 4 weeks) will be reported.
  The PROMIS assesses pain on a numeric rating scale from 0 (no pain) to 10 (worst imaginable pain)
Time Frame: Baseline, 2 weeks and 4 weeks
Population: Investigators discovered recently that there had been a protocol deviation such that a participant had had their surgery PRIOR to filling out the baseline survey. That participant's baseline data had to be removed from our analyses and revised data has been submitted. Not all participants provided evaluable data for analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group I eHealth Mindful Movement and Breathing (eMMB) | Group II Attention Control (AC)
Number analyzed (Participants) | 11 | 17
score on a scale
  Baseline | 3.63 (3.47) | 3.11 (3.41)
  2 weeks change in score: number analyzed (Participants) | 10 | 14
  2 weeks change in score | -1.9 (3.57) | -0.71 (2.67)
  4 weeks change in score: number analyzed (Participants) | 11 | 14
  4 weeks change in score | -2.55 (3.08) | -1.14 (3.03)

4. Secondary Outcome: Change in Affective Dimension of Pain
Description: The affective dimension of pain will be assessed with one item on a scale from 0 (not bad at all) to 10 (the most unpleasant feeling possible for me). A higher score represent a higher affective dimension of pain for the participant. A change in score between two or more time points (baseline, 2 weeks and 4 weeks) will be reported.
Time Frame: Baseline, 2 weeks and 4 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group I (eMMB) | Group II (AC)
Number analyzed (Participants) | 11 | 17
score on a scale
  Baseline | 3.09 (3.53) | 3.06 (3.75)
  2 weeks change in score: number analyzed (Participants) | 10 | 14
  2 weeks change in score | -1.00 (3.89) | -0.71 (3.67)
  4 weeks change in score: number analyzed (Participants) | 11 | 14
  4 weeks change in score | -2.00 (3.13) | -1.07 (2.92)

5. Secondary Outcome: Change in Pain Interference Per PROMIS Measure
Description: Baseline analyses will include descriptive statistics of pain, background characteristics and other possible confounding variables by intervention group. The primary goal of the statistical analysis of these measures for this Aim will be to estimate standard deviations (SD) for use in future studies. Additional analyses will include fitting mixed analysis of covariance (ANCOVA) models (adjustment for baseline) to model the trajectory of pain by time and group accounting for the repeated measures on a subject. Score range is 0-100 with a higher score representing greater pain interference for the participant. A change in score between two or more time points (baseline, 2 weeks and 4 weeks) will be reported.
Time Frame: Baseline, 2 weeks and 4 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group I (eMMB) | Group II (AC)
Number analyzed (Participants) | 11 | 17
score on a scale
  Baseline | 53.38 (11.22) | 55.02 (10.93)
  2 weeks change in score: number analyzed (Participants) | 10 | 14
  2 weeks change in score | -0.08 (13.88) | -0.93 (12.79)
  4 weeks change in score: number analyzed (Participants) | 11 | 14
  4 weeks change in score | -5.92 (10.82) | -4.00 (12.27)

6. Secondary Outcome: Change in Sleep Disturbances Per PROMIS Sleep Disturbance Short-form
Description: Baseline analyses will include descriptive statistics of pain, background characteristics and other possible confounding variables by intervention group. The primary goal of the statistical analysis of these measures for this Aim will be to estimate standard deviations (SD) for use in future studies. Score range is 0-100 with higher scores representing a greater sleep disturbance for participants. A change in score between two or more time points (baseline, 2 weeks and 4 weeks) will be reported.
Time Frame: Baseline, 2 weeks and 4 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group I (eMMB) | Group II (AC)
Number analyzed (Participants) | 11 | 17
score on a scale
  Baseline | 49.65 (11.78) | 52.46 (10.33)
  2 weeks change in score: number analyzed (Participants) | 10 | 14
  2 weeks change in score | -3.42 (9.03) | -2.92 (8.26)
  4 weeks change in score: number analyzed (Participants) | 11 | 14
  4 weeks change in score | -1.53 (8.15) | -1.90 (7.74)

7. Secondary Outcome: Change in Psychological Distress Per PROMIS Depression
Description: Baseline analyses will include descriptive statistics of pain, background characteristics and other possible confounding variables by intervention group. The primary goal of the statistical analysis of these measures for this Aim will be to estimate standard deviations (SD) for use in future studies. Score range is 0-100 with the higher score representing greater depression in the participants. A change in score between two or more time points (baseline, 2 weeks and 4 weeks) will be reported.
Time Frame: Baseline, 2 weeks and 4 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group I (eMMB) | Group II (AC)
Number analyzed (Participants) | 11 | 17
score on a scale
  Baseline | 51.43 (11.07) | 50.42 (8.51)
  2 weeks score change: number analyzed (Participants) | 10 | 14
  2 weeks score change | -7.38 (8.60) | -3.78 (9.98)
  4 weeks score change: number analyzed (Participants) | 11 | 14
  4 weeks score change | -6.58 (8.06) | -3.75 (5.47)

8. Secondary Outcome: Change in Psychological Distress Per PROMIS Anxiety
Description: Baseline analyses will include descriptive statistics of pain, background characteristics and other possible confounding variables by intervention group. The primary goal of the statistical analysis of these measures for this Aim will be to estimate standard deviations (SD) for use in future studies. Score range is 0-100 with a higher score presenting a greater level of anxiety in the participants. A change in score between two or more time points (baseline, 2 weeks and 4 weeks) will be reported.
Time Frame: Baseline, 2 weeks and 4 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group I (eMMB) | Group II (AC)
Number analyzed (Participants) | 11 | 17
score on a scale
  Baseline | 53.47 (12.29) | 55.49 (8.40)
  2 weeks change in score: number analyzed (Participants) | 10 | 14
  2 weeks change in score | -7.36 (7.83) | -9.66 (13.73)
  4 weeks change in score: number analyzed (Participants) | 11 | 14
  4 weeks change in score | -5.86 (9.70) | -7.90 (11.64)

9. Secondary Outcome: Incidence of Adverse Events Per Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0
Description: Will describe any adverse events reported as frequencies.
Time Frame: Up to 4 weeks
Measure: Number; unit: number of adverse events
Arm/Group | Group I (eMMB) | Group II (AC)
Number analyzed (Participants) | 11 | 14
number of adverse events | 0 | 0

ADVERSE EVENTS:
Time Frame: Four weeks
Arm/Group | Group I (eMMB) | Group II (AC)
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/17
Other Adverse Events (participants affected / at risk) | 0/13 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-08-19): https://cdn.clinicaltrials.gov/large-docs/05/NCT03681405/Prot_SAP_000.pdf
  • Informed Consent Form (2019-09-09): https://cdn.clinicaltrials.gov/large-docs/05/NCT03681405/ICF_001.pdf